CLINICAL TRIAL: NCT02605915
Title: A Phase Ib, Open-Label Study Evaluating the Safety and Pharmacokinetics of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Trastuzumab Emtansine or With Trastuzumab and Pertuzumab (With and Without Docetaxel) in Patients With HER2-Positive Breast Cancer and Atezolizumab With Doxorubicin and Cyclophosphamide in HER2-Negative Breast Cancer
Brief Title: Safety and Pharmacokinetics of Atezolizumab Combination Treatments in Participants With HER2-Positive and HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29831; 2015-002113-29 (EudraCT Number)
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: HER2-Positive Metastatic Breast Cancer; HER2-Negative Metastatic Breast Cancer; Locally Advanced or Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Carboplatin; Docetaxel; pertuzumab; Trastuzumab; Ado-Trastuzumab Emtansine; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1A: Atezolizumab/Trastuzumab/Pertuzumab (Experimental): Participants will receive atezolizumab in combination with trastuzumab and pertuzumab every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 1B: Atezolizumab/Trastuzumab emtansine 3.6 mg (Experimental): Participants will receive atezolizumab in combination with trastuzumab emtansine (3.6 mg/kg) every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab emtansine
- Cohort 1C: Atezolizumab/Trastuzumab emtansine 3.0 mg (Experimental): Participants will receive atezolimumab in combination with trastzumab emtansine (3.0 mg/kg) every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab emtansine
- Cohort 1D: Atezolizumab/Trastuzumab emtansine 2.4 mg (Experimental): Participants will receive atezolimumab in combination with trastzumab emtansine (2.4 mg/kg) every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab emtansine
- Cohort 1E: Atezolizumab/ doxorubicin/ cyclophosphamide (Experimental): Participants with HER2-negative breast cancer will receive atezolizumab (every 2 weeks) in combination with doxorubicin (every 2 weeks) and cyclophosphamide for four cycles. After the completion of four cycles of combination atezolizumab /doxorubicin / cyclophosphamide, atezolizumab will be continued as a single-agent at a dose of 1200 mg every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide
- Cohort 1F: Atezolizumab/Trastuzumab/Pertuzumab/ Docetaxel (Experimental): Participants will receive atezolizumab in combination with trastuzumab, pertuzumab, and docetaxel every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 2A: Atezolizumab/Trastuzumab/Pertuzumab (Experimental): Participants will receive atezolizumab in combination with trastuzumab and pertuzumab every 3 weeks for 2 cycles, followed by docetaxel, carboplatin, trastuzumab and pertuzumab every 3 weeks for 6 cycles. Breast surgery will be performed no later than 6 weeks after neoadjuvant therapy. Upon the completion of surgery, participants will receive 12 cycles of single-agent trastuzumab every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 2B: Atezolizumab/Trastuzumab emtansine (Experimental): Participants will receive atezolizumab in combination with trastuzumab emtansine every 3 weeks for 2 cycles, followed by docetaxel, carboplatin, trastuzumab and pertuzumab every 3 weeks for 6 cycles. Breast surgery will be performed no later than 6 weeks after neoadjuvant therapy. Upon the completion of surgery, participants will receive 12 cycles of single-agent trastuzumab every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab; Drug: Trastuzumab emtansine
- Cohort 2C: Safety Expansion (Experimental): Participants with HER2-positive metastatic breast cancer/unresectable locally advanced breast cancer who received prior treatment with trastuzumab and a taxane chemotherapy will receive atezolizumab in combination with trastuzumab emtansine at the dose determined from stage 1, every 3 weeks until disease progression, lack of clinical benefit, or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab emtansine
- Cohort 2D: Safety Expansion (Experimental): Participants with HER2-positive metastatic breast cancer recently progressed on an HP containing regimen will receive atezolimumab in combination with trastuzumab and pertuzumab every 3 weeks until disease progression, lack of clinical benefit, or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 milligrams (mg) or 840 mg (Cohort 1E only) flat dose administered via intravenous (IV) infusion on Day 1 of every 21-day cycle.
  Other Names: Tecentriq, RO5541267
Drug: Carboplatin — Carboplatin will be administered at an initial target of area under the curve (AUC) of 6 milligrams per milliliter*min (mg/mL*min) via an IV infusion on Day 1 of every 21-days for 6 cycles.
  Arms: Cohort 2A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 2B: Atezolizumab/Trastuzumab emtansine
Drug: Docetaxel — Docetaxel 75 mg/m^2 administered via IV infusion on Day 1 every 21-days for 6 cycles.
  Arms: Cohort 1F: Atezolizumab/Trastuzumab/Pertuzumab/ Docetaxel; Cohort 2A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 2B: Atezolizumab/Trastuzumab emtansine
Drug: Pertuzumab — Pertuzumab 840 mg loading dose then 420 mg administered via IV infusion on Day 1 of every 21-day cycle.
  Other Names: RO4368451
  Arms: Cohort 1A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 1F: Atezolizumab/Trastuzumab/Pertuzumab/ Docetaxel; Cohort 2A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 2B: Atezolizumab/Trastuzumab emtansine; Cohort 2D: Safety Expansion
Drug: Trastuzumab — Trastuzumab 8 milligram per kilogram (mg/kg) loading dose, then 6 mg/kg administered via IV infusion on Day 1 of every 21-day cycle.
  Other Names: RO0452317
  Arms: Cohort 1A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 1F: Atezolizumab/Trastuzumab/Pertuzumab/ Docetaxel; Cohort 2A: Atezolizumab/Trastuzumab/Pertuzumab; Cohort 2B: Atezolizumab/Trastuzumab emtansine; Cohort 2D: Safety Expansion
Drug: Trastuzumab emtansine — Trastuzumab emtansine 3.6 mg/kg administered via IV infusion on Day 1 of every 21-day cycle. Dose de-escalation may occur for trastuzumab emtansine, from the full trastuzumab emtansine dose at 3.6 mg/kg on Day 1 of every 21-day cycle, potentially to 3.0 mg/kg (Cohort 1C) or 2.4 mg/kg q3w (Cohort 1D).
  Other Names: RO5304020
  Arms: Cohort 1B: Atezolizumab/Trastuzumab emtansine 3.6 mg; Cohort 1C: Atezolizumab/Trastuzumab emtansine 3.0 mg; Cohort 1D: Atezolizumab/Trastuzumab emtansine 2.4 mg; Cohort 2B: Atezolizumab/Trastuzumab emtansine; Cohort 2C: Safety Expansion
Drug: Doxorubicin — Doxorubicin will be administered at 60 mg/m^2 every 2 weeks as an IV bolus over 3 to 5 minutes or as an infusion over 15 to 30 minutes.
  Arms: Cohort 1E: Atezolizumab/ doxorubicin/ cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 600 mg/m^2 on Day 1 of each 21 day cycle as an IV bolus over 3 to 5 minutes or as an infusion, in accordance with local policy.
  Arms: Cohort 1E: Atezolizumab/ doxorubicin/ cyclophosphamide

SUMMARY:
This is a Phase Ib, open-label, two-stage study with two active regimens in each stage designed to evaluate the safety and tolerability of combination treatment with atezolizumab, trastuzumab, and pertuzumab (with and without docetaxel) or atezolizumab and trastuzumab emtansine in participants with human epidermal growth factor receptor 2 (HER2) positive metastatic breast cancer (MBC) and locally advanced early breast cancer (EBC), and atezolizumab with doxorubicin and cyclophosphamide in HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented HER2-positive and HER2-negative (cohort E only) breast cancer
* Metastatic breast cancer that is measurable (Stage 1) or early breast cancer with a primary tumor size greater than (>) 2 centimeter (cm) (Stage 2)
* Eastern cooperative oncology group (ECOG) performed status of 0, 1 or 2; 0 or 1 (cohort E only)
* Life expectancy of 12 or more weeks
* Adequate hematologic and end-organ function
* Left ventricular ejection fraction greater than or equal to (>=) 50 percentage (%); >=55% (cohort E only)

Exclusion Criteria:

* Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases
* Leptomeningeal disease
* Pregnancy or lactation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2015-12-31 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities (DLT) - Cohort 1A, 1B, 1C, 1D, 1F | Baseline up to Day 21
Percentage of Participants With DLT - Cohort 1E | Baseline up to Day 28
Percentage of Participants With Adverse Events (AEs) According to National Cancer Institute Common Terminology Criteria for AEs, Version 4.0 (NCI CTCAE V4.0) | Baseline up to approximately 3 years

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Atezolizumab | Cohorts 1A, 1B, 1C, 1D, E1, 1F, 2A, 2B, 2C, 2D: pre-infusion (Hour 0), 30 minutes after end of atezolimumab infusion on Day 1 Cycle 1 (cycle length=21 days) up to approximately 3 years (detailed timeframe provided in measure description)
  Cohorts 1A, 1B, 1C, 1D, E1, 1F, 2A, 2B, 2C, 2D: 30 minutes after end of infusion on Day 1 Cycle 1 (cycle length=21 days); pre-infusion (Hour 0) on Day 1 of Cycle 1, 2, 3 (except cohort 1E), 4, 8, on Day 1 of every 8 cycles until study treatment/early discontinuation, 120 days after treatment completion/discontinuation (up to approximately 3 years)
Minimum Serum Concentration (Cmin) of Atezolizumab | pre-infusion (Hour 0) on Day 1 of Cycle 1, 2, 3 (except cohort 1E), 4, 8 (cycle length=21 days), on Day 1 of every 8 cycles until study treatment/early discontinuation, 120 days after treatment completion/discontinuation (up to approximately 3 years)
Cmin of Trastuzumab | Cohorts 1A, 1F, 2A, 2D: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Cmin of Trastuzumab Emtansine | Cohorts 1B, 1C, 1D, 2B, 2C: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Cmin of Pertuzumab | Cohorts 1A, 1F, 2A, 2D: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Cmin of Doxorubicin | Cohort 1E: at the end of doxorubicin infusion, 4 and 8 hours after doxorubicin infusion on Day 1 of Cycle 1 and 4 (cycle length=21 days)
Cmin of Cyclophosphamide | Cohort 1E: at the end of cyclophosphamide infusion on Day 1 of Cycle 1 and 4 (cycle length=21 days), 4 and 8 hours after cyclophosphamide infusion on Day 1 of Cycle 1
Percentage of Participants With Anti-Therapeutic Antibody (ATA) Response to Atezolimumab | pre-infusion (Hour 0) on Day 1 of Cycle 1, 2, 3 (except cohort 1E), 4, 8 (cycle length=21 days), on Day 1 of every 8 cycles until study treatment/early discontinuation, 120 days after treatment completion/discontinuation (up to approximately 3 years)
Percentage of Participants With Anti-Therapeutic Antibody (ATA) Response to Trastuzumab | Cohorts 1A, 1F, 2A, 2D: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Percentage of Participants With Anti-Therapeutic Antibody (ATA) Response to Trastuzumab Emtansine | Cohorts 1B, 1C, 1D, 2B, 2C: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Percentage of Participants With Anti-Therapeutic Antibody (ATA) Response to Pertuzumab | Cohorts 1A, 1F, 2A, 2D: pre-infusion (Hour 0) on Day 1 of Cycle 1, 3 (cycle length=21 days), at study treatment/early discontinuation, 120 days after treatment completion or discontinuation (up to approximately 3 years)
Number of Treatment Cycles Received | Baseline up to approximately 3 years
Percentage of Participants With Various Dose Intensity | Baseline up to approximately 3 year
Plasma Concentration of Doxorubicin | Cohort 1E: at the end of doxorubicin infusion, 4 and 8 hours after doxorubicin infusion on Day 1 Cycle 1 and 4 (cycle length=21 days)
Plasma Concentration of Cyclophosphamide | Cohort 1E: at the end of cyclophosphamide infusion on Day 1 of Cycle 1 and 4 (cycle length=21 days), 4 and 8 hours after cyclophosphamide infusion on Day of Cycle 1
Plasma Concentration of 4-Hydroxycyclophosphamide | Cohort 1E: at the end of cyclophosphamide infusion on Day 1 of Cycle 1 and 4 (cycle length=21 days), 4 and 8 hours after cyclophosphamide infusion on Day of Cycle 1
Plasma Concentration of Docetaxel | Cohort 1F: at the end of docetaxel infusion, 4 and 8 hours after docetaxel infusion on Day 1 Cycle 1 and 3 (cycle length=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences; Winthrop Rockefeller Cancer Institute, Little Rock, Arkansas
  - Joliet oncology hematology associates, Joliet, Illinois
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Karmanos Cancer Center; Department of Oncology, Detroit, Michigan
  - HCA Midwest Division, Kansas City, Missouri
  - Montefiore Medical Center, Advanced Women's Health Center, Clinical Trials and Research Unit; Depart, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology - Chattanooga; Tennessee Oncology - East Third Street, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center CTRC at UTHSCSA, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin